CLINICAL TRIAL: NCT00165074
Title: Pilot Trial of Surfactant Therapy For Preterm Neonates 5-21 Days Old With
Brief Title: Pilot Trial of Surfactant Therapy For Preterm Neonates 5-21 Days Old With Respiratory Decompensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Women & Children's Hospital of Buffalo (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002-9-2968
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Respiratory Distress Syndrome
Keywords: Prematurity; Lung Disease; Hyaline Membrane; Surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth; Lung Diseases | interventions — calfactant; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Infasurf (drug) — Infasurf 3 cc/kg instilled via endotracheal tube q 12-24 hours x 2 doses
  Other Names: Infasurf (calfactant, manufactured for Forest Pharmaceuticals, Inc. St. Louis, MO, by ONY Inc., Amherst, NY

SUMMARY:
The purpose of the study is to determine whether additional surfactant(Infasurf) doses at 7 to 10 days of life time will improve lung function in premature infants, allowing a decrease in required oxygen concentration and ventilator settings.

DETAILED DESCRIPTION:
Pulmonary surfactant is required for normal lung function. Preliminary data from previous trials suggest that more than half of chronically ventilated premature infants, greater than 1 week of age, have at least one episode of surfactant dysfunction, as measured in vitro, associated with a low surfactant protein B content. We propose to enroll premature infants less than 1250 gm birthweight, between days 5 and 21 of life who are intubated, mechanically ventilated, with a respiratory decompensation, defined as a severity score (mean airway pressure x FIO2) rising from a baseline of < 1.8 to > 3.5, sustained for > 24 hours. Infants will receive two doses of Infasurf surfactant, 12-24 hours apart, at the standard dose of 3 ml/kg. Primary outcome is the change in respiratory severity score at 72 hours post surfactant treatment compared to pre-treatment. Sample size is 31 infants, study duration is 3 years, and recruitment of study patients will occur at the Hospital of the University of Pennsylvania, and Women and Children's Hospital of Buffalo.

ELIGIBILITY:
Inclusion Criteria:

* Less than 1250 gm birthweight
* Day 5-21 of life
* Intubated and mechanically ventilated, with respiratory decompensation, defined as the majority of daily severity scores (calculated every 6 hr from average of respiratory settings over 3-4 hour period) rising from baseline < 1.8, to > 3.5, sustained for >24hr. Note: Prior surfactant therapy at birth is neither an inclusion nor exclusion criterion.

Exclusion Criteria:

* Serious congenital malformations
* Life expectancy < 7 days from enrollment
* Patent ductus arteriosus at time of decompensation
* Pulmonary hemorrhage as cause of respiratory decompensation
* Active air leak syndrome at time of decompensation
* Postnatal steroid therapy for lung disease

Ages: 7 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2003-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
We hypothesize that at least 25% of treated infants will have a 50% or greater reduction in respiratory severity score at 72 hours compared to pre-treat | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Posencheg, MD, Principal Investigator — University of Pennsylvania/Children's Hospital of Philadelphia; Roberta A Ballard, MD, Principal Investigator — University of California, San Francisco Medical Center

REFERENCES:
- [Background] Merrill JD, Ballard RA, Cnaan A, Hibbs AM, Godinez RI, Godinez MH, Truog WE, Ballard PL. Dysfunction of pulmonary surfactant in chronically ventilated premature infants. Pediatr Res. 2004 Dec;56(6):918-26. doi: 10.1203/01.PDR.0000145565.45490.D9. Epub 2004 Oct 20. PMID 15496605